CLINICAL TRIAL: NCT06086509
Title: Effect of Music on Fear and Anxiety in Children During Tomography: Randomized Controlled Double-Blind Study
Brief Title: Letting Children Listen to Music During Computed Tomography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gümüşhane Universıty (Other)
Responsible Party: Principal Investigator, Zeynep Demir, lecturer, Gümüşhane Universıty
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: A/BU-HEM-ZDİ-01
Record Dates: First submitted 2023-09-30; First posted 2023-10-17 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Fear; Computed Tomography
Keywords: Child; Music; Anxiety; Fear
MeSH Terms: conditions — Anxiety Disorders | interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: They were divided into two groups: control group and experimental group.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blindness method was used to avoid bias in this study. The researcher, who evaluated the children's anxiety and fear levels during and after the tomography in order to prevent selection bias, did not know which group the children and their families were in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): Questionnaires and scales were filled out by the researcher five minutes before the CT scan. Routine CT scans were performed on the control group without listening to music by wearing a Bluetooth headset. The scales were repeated five minutes after the CT scan.
- music group (Experimental): Questionnaires and scales were filled out by the researcher five minutes before the CT scan. Just before the CT scan began, the children in the music group were started to listen to "Lullaby K 350" music by inserting a Bluetooth headset into their ears. If the process took longer, the music was played again. Additionally, the Bluetooth headset was properly disinfected before each use to prevent the spread of infectious diseases among patients.
  Interventions: Other: Music

INTERVENTIONS:
Other: Music — Children were played music during computerized tomography.
  Arms: music group

SUMMARY:
This study examines the effect of music during computed tomography in children. This study, conducted on a total of 60 children, was divided into two groups: the music group and the control group. According to the research results; showed that music reduces fear and anxiety levels in children and stabilizes vital signs (pulse and respiratory rate) during a tomography scan.

DETAILED DESCRIPTION:
Aim: This research was conducted to determine the effect of music played during computerized tomography (CT) imaging in children on fear, anxiety and vital signs.

Method: This randomized, double-blind controlled trial was conducted with Consolidated Standards of Reporting Studies (CONSORT) guidelines. The sample includes children aged 5-10 years who had CT scans in the emergency department of a public hospital in eastern Turkey between April 18 and May 20, 2023 and met the inclusion criteria for the study. The research was completed with a total of 60 children, divided evenly into one of two groups. The nursing intervention of the research is to listen to music. Data were collected through face-to-face interviews using the Child and Family Information Form, the Child Fear Scale, the State Anxiety Scale for Children, and the Vital Signs Monitoring Form (pulse, blood pressure, and oxygen saturation). Ethical principles were followed in the research.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 5-10
* Hospitalization is for diagnostic or treatment purposes
* The child and the parent speak and understand Turkish comfortably.

Exclusion Criteria:

* Having previous tomography shooting experience
* Having chronic diseases
* Visual, auditory, speech and mental disorders
* There is a history of sedative, analgesic or narcotic substance use within 24 hours before application.

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2023-04-18 (Actual); Primary Completion 2023-05-20 (Actual); Study Completion 2023-09-20 (Actual)

PRIMARY OUTCOMES:
Children's Fear Scale (CFS) | one month
  Children's Fear Scale is a scale scored between 0 and 4 showing five faces varying between a neutral expression (0 = no fear) to fearful face (4 = extreme fear).

SECONDARY OUTCOMES:
Child Anxiety Scale-State (CAS-S) | one month
  The Child Anxiety Scale-State Scale resembles a thermometer with a bulb at the bottom and horizontal lines at intervals going upwards. This scale, for children ages 4 to 10, instructs children to "Imagine that all your anxious or nervous feelings are in the bulb or bottom part of the thermometer

CONTACTS AND LOCATIONS:
Overall Officials: Fatma KURUDİREK, Principal Investigator — Ataturk University
Locations (1):
- Gümüşhane University, Gümüşhane, Turkey (Türkiye)

REFERENCES:
- [Derived] Kurudirek F, Demir Barbak Z, Demir Imamoglu Z, Ciftci K, Delice O. The Effect of Music on Fear and Anxiety of Children During Tomography: A Randomized Controlled Double-Blind Study. Int J Nurs Pract. 2025 Jun;31(3):e70029. doi: 10.1111/ijn.70029. PMID 40511812